CLINICAL TRIAL: NCT02896972
Title: Efficacy of Inverted Internal Limiting Membrane Flap Technique for Macular Hole Retinal Detachment in Highly Myopic Eyes
Brief Title: Inverted Internal Limiting Membrane Flap Technique for Macular Hole Retinal Detachment in Highly Myopic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Professor of Ophthalmology, Kyorin University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kyorineye022
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Macular Hole Retinal Detachment
Keywords: vitrectomy; macular hole retinal detachment; high myopia
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inverted ILM flap group (Active Comparator): Eyes underwent vitrectomy with inverted internal limiting membrane technique
  Interventions: Procedure: Vitrectomy
- ILM peeling group (Active Comparator): Eyes underwent vitrectomy with internal limiting membrane peeling
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy — Vitrectomy with inverted ILM technique or ILM peeling

SUMMARY:
To evaluate efficacy of vitrectomy with inverted internal limiting membrane (ILM) flap technique for macular hole retinal detachment (MHRD) in highly myopic eyes, and to demonstrate postoperative clinical course of MHRD after inverted ILM flap technique using swept-source optical coherence tomography (OCT)

DETAILED DESCRIPTION:
Macular hole retinal detachment (MHRD) threatens a certain number of highly myopic patients for irreversible visual dysfunction, and mostly requires immediate surgical intervention. The aim of they study is to evaluate efficacy of vitrectomy with inverted internal limiting membrane (ILM) flap technique for MHRD in highly myopic eyes, and to demonstrate postoperative clinical course of MHRD after inverted ILM flap technique using swept-source optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients who underwent vitrectomy and internal limiting membrane removal or inverted for macular hole retinal detachment and had followed for more than 6 months.

Exclusion Criteria:

* The patients with follow-up less than 6 months.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Visual acuity before and after surgery | Changes from baseline to 1, 3, 6 months

SECONDARY OUTCOMES:
Optical coherence tomography | Changes from baseline up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center

IPD SHARING:
Plan to Share IPD: Undecided